CLINICAL TRIAL: NCT03134378
Title: Comparison of Triple Therapy Regimens Effectiveness Over 10 Days and 14 Days in Eradication of Helicobacter Pylori Infection: Double Blind Randomized Clinical Trial
Brief Title: 10 vs 14 Days Triple Therapy : H.Pylori Infection Eradication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ari Fahrial Syam, Dr. dr. SpPD, K-GEH, MMB, FACP, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-10-311
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; triple therapy; eradication
MeSH Terms: interventions — Rabeprazole; Clarithromycin; Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized-double blinded Clinical Trials
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 14 days triple therapy (Experimental): Rabeprazole Clarithromycin Amoxicillin
  Interventions: Drug: Rabeprazole Sodium 20mg; Drug: Clarithromycin 500mg; Drug: Amoxicillin 500 Mg
- 10 days triple therapy (Placebo Comparator): Rabeprazole Clarithromycin Amoxicillin
  Interventions: Drug: Rabeprazole Sodium 20mg; Drug: Clarithromycin 500mg; Drug: Amoxicillin 500 Mg

INTERVENTIONS:
Drug: Rabeprazole Sodium 20mg — Twice daily
  Other Names: Pariet
Drug: Clarithromycin 500mg — Twice daily
  Other Names: Bicrolid
Drug: Amoxicillin 500 Mg — Twice daily
  Other Names: Amoxicillin generic

SUMMARY:
Helicobacter pylori is a bacterium estimated to colonize in the gastrointestinal tract of the half population in the world. Colonization of this bacteria is suspected to be one of the main risk factor for the occurrence of various abnormalities of the upper gastrointestinal tract, such as peptic ulcer and gastrointestinal cancer. The Experts recommend giving triple therapy regimens as first-line eradication therapy for Helicobacter pylori infection. The recommended duration of triple therapy is 10-14 days. However, recent studies suggest triple therapy with longer duration will provide a higher percentage of eradication. This study wanted to show whether 14 days of triple therapy was better than 10 days in Helicobacter pylori eradication.

DETAILED DESCRIPTION:
This is a double-blinded randomized clinical trials, to determine the proportion of eradication of Helicobacter pylori infection using a triple therapy regimen for 10 days and 14 days. The triple therapy regimen was a proton pump inhibitor (Rabeprazole 20 mg twice daily), Amoxicillin 1000 mg twice daily, and Clarithromycin 500 mg twice daily.

Patients with dyspepsia and no improvement for at least 2 weeks with empiric therapy (lifestyle education, antacid, H2-antagonist, or proton pump inhibitor), are further investigated to determine the presence of Helicobacter pylori infection using invasive (Esophagoduodenoscopy/EGD) or non-invasive methods (Urea Breath Test/UBT).

Patients with positive results on UBT or histology examination from EGD and fulfill inclusion and exclusion criteria are included as research subjects, then randomly assigned to determine the subject of the study into the sample of study entry in group 1 or group 2.

All subjects will be required to fill out informed consent, demographic data, anthropometric measurements, and questionnaires.

Research subjects will get triple therapy regimen for Helicobacter pylori infection in the form of Proton Pump Inhibitor (Rabeprazole 2 x 20 mg), Amoxicillin 2 x 1000 mg, and Clarithromycin 2 x 500 mg.

Pharmacy will create two sets of regimens, in which one group of regimens contains triple therapy regimens for 10 days followed by the same regimen for 4 days, while another regimen group contains triple therapy regimens for 10 days Day followed by placebo for 4 days. Neither the researcher nor the study subjects knew the triple therapy regimen given to group 1 and group 2 subjects, and only became known after the end of the study.

All subjects will be monitored given drug consumption and evaluated regularity, complaints, and adverse effects arising for 14 days by researchers. The patient is given a control card to write down medication time and any possible complaints or side effects of drug allergic reactions, epigastric pain, headache, discomfort, and nausea / vomiting, and other side effects will be observed during the study. The patient will be determined whether the study will continue or not.

After the therapy was completed, the subjects of the study will be re-examined as an evaluation of eradication success, at least 28 days after completion of triple therapy regimen.

If UBT negative results obtained at the time of evaluation, the eradication is success, when positive UBT results are obtained at the time of evaluation, eradication is failed and the subjects are persistent with first-line therapy.

Persistent patients are encouraged to undergo an EGD at Cipto Mangunkusumo Hospital for the culture of Helicobacter pylori infection resistance. If the patient is not willing to be underwent EGD, then the patient is given second-line treatment regimen of Levofloxacin 2 x 500 mg, Amoxicillin 2 x 1000 mg, and Rabeprazole 2 x 20mg.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older patients who are proven to be infected by Helicobacter pylori based on positive in Urea Breath Test or positive in histopathologic examination of biopsy in antrum and corpus of gaster through esophagoduodenoscopy.

Exclusion Criteria:

* Patients refuse to follow the research
* Patient has had previous eradication therapy of Helicobacter pylori infection.
* The patient is pregnant or breastfeeding
* Patients have a history of allergy to one component of triple therapy regimen (proton pump inhibitor, penicillin, and / or macrolide) before.
* Patients are known to have impaired liver function, evidenced by ALT values within normal limits, and no previous liver disease.
* Patients were found to have arrhythmias or obtained QT wave elongation on electrocardiographic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2016-10-03 (Actual); Primary Completion 2017-05-05 (Estimated); Study Completion 2017-05-12 (Estimated)

PRIMARY OUTCOMES:
Eradication of Helicobacter pylori infection | 4 weeks after completed therapy
  Urea Breath Test after therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No